CLINICAL TRIAL: NCT02896205
Title: A Randomized Controlled Trial to Compare the Efficacy of Oral Mycophenolate Mofetil With Placebo in Patients With Systemic Sclerosis Related Early Interstitial Lung Disease
Brief Title: Study to Compare the Efficacy of Mycophenolate Mofetil in Systemic Sclerosis Related Early Interstitial Lung Disease
Acronym: MYILD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, GSRSNK NAIDU, SENIOR RESIDENT, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NK/2612/DM/10772
Record Dates: First submitted 2016-08-27; First posted 2016-09-12 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Systemic Sclerosis; Scleroderma; Interstitial Lung Disease
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Lung Diseases, Interstitial | interventions — Mycophenolic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mycophenolate mofetil (Experimental): Subjects will be started on Mycophenolate Mofetil 500mg twice a day and increased by 500mg every 2 weeks, if tolerated, to a target dose of 2gram per day.
  Interventions: Drug: Mycophenolate mofetil
- Placebo (Placebo Comparator): Subjects in this arm will be given matching placebo, made of lactulose, starting at two tablets per day and increased by one tablet every 2 weeks to a target of 4 tablets per day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mycophenolate mofetil — Subjects will be given oral Mycophenolate Mofetil starting at 500mg twice a day and increased gradually to a target dose of 2gram per day for 6 months
  Other Names: MMF
  Arms: Mycophenolate mofetil
Drug: Placebo — Subjects will be given matching placebo for 6 months
  Arms: Placebo

SUMMARY:
Systemic sclerosis is a multisystem disease and can involve the lungs in the form of ILD. Lung involvement is the most common cause of death in these patients. The present study is performed to study the efficacy of oral mycophenolate mofetil in treating early and mild ILD in patients of SSc. The efficacy and side effects of mycophenolate mofetil will be compared with that of oral placebo.

DETAILED DESCRIPTION:
Lung involvement is the leading cause of death among patients with systemic sclerosis (SSc). Treatment with immunosuppression drugs helps in retarding the progression of interstitial lung disease (ILD) and improves the morbidity and mortality among these patients. Presently, cyclophosphamide has been shown to be useful in stabilizing the lung functions among patients of systemic sclerosis with ILD. But use of cyclophosphamide is also associated with many adverse effects including infections, cytopenias, gonadal dysfunction and malignancies. Use of oral mycophenolate mofetil (MMF) in SSc-ILD in recent studies has been shown to be effective in retarding progression of ILD among these patients with a better side effect profile compared to cyclophosphamide. Contemporary expert opinion dictates that the treatment for SSc-ILD needs to be individualized. Generally, intense immunosuppression is required in patients with FVC <70% of the predicted. In patients with FVC >70% of the predicted, the need for high dose immunosuppression is not clear and varies from center-to-center. The present study is designed to determine the efficacy of oral MMF in patients with SSc related early ILD. The subjects in this study will be given either oral MMF or placebo and will be monitored for their response and adverse events. Informed consent will be taken from the subjects before including in the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients of systemic sclerosis with presence of interstitial lung disease on High Resolution Computer Tomography (HRCT) chest
2. FVC ≥ 70% of predicted on pulmonary function tests
3. Age ≥18 years
4. Consenting for participating in study

Exclusion Criteria:

1. Received immunosuppression (except low dose steroids, prednisolone equivalent ≤10 mg/day) for ILD in the last 3 years
2. Persistent leucopenia or thrombocytopenia
3. Pregnant or breastfeeding females
4. Severe pulmonary arterial hypertension (mean pulmonary arterial pressure >55mmHg) requiring drug therapy
5. Uncontrolled congestive heart failure
6. Any other abnormalities noted on chest X-ray or HRCT other than ILD
7. Active infection
8. Inflammatory myositis
9. Overlap syndrome
10. Mixed connective tissue disease
11. Other serious co-morbidities which could compromise patient's ability to complete the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2016-10; Primary Completion 2017-07-01 (Actual); Study Completion 2017-07-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Forced vital capacity (FVC) at 6 months, after treatment with oral mycophenolate mofetil or placebo | 6 months

SECONDARY OUTCOMES:
Change from baseline in Quality of Life (QoL) score by Medical Outcome Short Form 36 (SF-36v2) at 6 months | 6 months
Change from baseline in Mahler Dyspnoea Index (MDI) at 6 months | 6 months
Number of participants with serious and non seroius adverse events with mycophenolate mofetil (MMF) and placebo | 6 months
Change in Forced Vital Capacity (FVC) from baseline to 6 months according to antibody (anti-centromere and anti-topoisomerase1) profile | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: GSRSNK Naidu, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- PGIMER, Chandigarh, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tashkin DP, Elashoff R, Clements PJ, Goldin J, Roth MD, Furst DE, Arriola E, Silver R, Strange C, Bolster M, Seibold JR, Riley DJ, Hsu VM, Varga J, Schraufnagel DE, Theodore A, Simms R, Wise R, Wigley F, White B, Steen V, Read C, Mayes M, Parsley E, Mubarak K, Connolly MK, Golden J, Olman M, Fessler B, Rothfield N, Metersky M; Scleroderma Lung Study Research Group. Cyclophosphamide versus placebo in scleroderma lung disease. N Engl J Med. 2006 Jun 22;354(25):2655-66. doi: 10.1056/NEJMoa055120. PMID 16790698
- [Background] Hoyles RK, Ellis RW, Wellsbury J, Lees B, Newlands P, Goh NS, Roberts C, Desai S, Herrick AL, McHugh NJ, Foley NM, Pearson SB, Emery P, Veale DJ, Denton CP, Wells AU, Black CM, du Bois RM. A multicenter, prospective, randomized, double-blind, placebo-controlled trial of corticosteroids and intravenous cyclophosphamide followed by oral azathioprine for the treatment of pulmonary fibrosis in scleroderma. Arthritis Rheum. 2006 Dec;54(12):3962-70. doi: 10.1002/art.22204. PMID 17133610
- [Background] Tashkin DP, Roth MD, Clements PJ, Furst DE, Khanna D, Kleerup EC, Goldin J, Arriola E, Volkmann ER, Kafaja S, Silver R, Steen V, Strange C, Wise R, Wigley F, Mayes M, Riley DJ, Hussain S, Assassi S, Hsu VM, Patel B, Phillips K, Martinez F, Golden J, Connolly MK, Varga J, Dematte J, Hinchcliff ME, Fischer A, Swigris J, Meehan R, Theodore A, Simms R, Volkov S, Schraufnagel DE, Scholand MB, Frech T, Molitor JA, Highland K, Read CA, Fritzler MJ, Kim GHJ, Tseng CH, Elashoff RM; Sclerodema Lung Study II Investigators. Mycophenolate mofetil versus oral cyclophosphamide in scleroderma-related interstitial lung disease (SLS II): a randomised controlled, double-blind, parallel group trial. Lancet Respir Med. 2016 Sep;4(9):708-719. doi: 10.1016/S2213-2600(16)30152-7. Epub 2016 Jul 25. PMID 27469583
- [Derived] Naidu GSRSNK, Sharma SK, Adarsh MB, Dhir V, Sinha A, Dhooria S, Jain S. Effect of mycophenolate mofetil (MMF) on systemic sclerosis-related interstitial lung disease with mildly impaired lung function: a double-blind, placebo-controlled, randomized trial. Rheumatol Int. 2020 Feb;40(2):207-216. doi: 10.1007/s00296-019-04481-8. Epub 2019 Dec 7. PMID 31813058